CLINICAL TRIAL: NCT06395818
Title: The Effectiveness of Hyaluronic Acid on Prefabricated CAD CAM Bone Blocks for Ridge Augmentation: A Split Mouth Study
Brief Title: the Effect of Hyaluronic Acid on a Prefabricated CAD-CAM Bone Blocks for Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Helal, lecturer of oral medicine, periodontology, oral diagnosis and radiology department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6789
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Atrophy of Edentulous Alveolar Ridge
Keywords: CAD-CAM bone blocks; hyaluronic acid; histomorphometric analysis

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: using closed envelop for participants the data will be given to outcomes assessors without defining the intervention for each group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prefabricated CAD-CAM allogeneic bone block hydrated using hyaluronic acid (Experimental): mucoperiosteal flap will be elevated to expose the atrophic ridge then the prefabricated CAD-CAM allogenic block will be fixed in its position with titanium miniscrews , The block was coated with a nonporous d-PTFE membrane
  Interventions: Procedure: prefabricated CAD-CAM allogeneic bone block hydrated using hyaluronic acid
- prefabricated CAD-CAM allogeneic bone block sterilized hydrated using saline solution (Experimental): mucoperiosteal flap will be elevated to expose the atrophic ridge then the prefabricated CAD-CAM allogenic block will be fixed in its position with titanium miniscrews ,The block was coated with a nonporous d-PTFE membrane
  Interventions: Procedure: prefabricated CAD-CAM allogeneic bone block sterilized hydrated using saline solution

INTERVENTIONS:
Procedure: prefabricated CAD-CAM allogeneic bone block hydrated using hyaluronic acid — exposure of atrophic posterior mandibular ridge, augmentation with CAD-CAM prefabricated allogenic bone block which fixed with titanium screws ,The block was coated with a nonporous d-PTFE membrane
  Arms: prefabricated CAD-CAM allogeneic bone block hydrated using hyaluronic acid
Procedure: prefabricated CAD-CAM allogeneic bone block sterilized hydrated using saline solution — exposure of atrophic posterior mandibular ridge, augmentation with CAD-CAM prefabricated allogenic bone block which fixed with titanium screws. The block was coated with a nonporous d-PTFE membrane
  Arms: prefabricated CAD-CAM allogeneic bone block sterilized hydrated using saline solution

SUMMARY:
Each patient will receive 2 prefabricated CAD-CAM allogeneic bone blocks sterilized with gamma rays with different rehydration methods.

Side I: prefabricated CAD-CAM allogeneic bone block sterilized with gamma rays hydrated using hyaluronic acid * Side II: prefabricated CAD-CAM allogeneic bone block sterilized with gamma rays hydrated using saline solution Both blocks are fixed with osteosynthesis screws, covered with non resorbable membranes** The membranes will be removed after 6 months, dental implants will be placed and core biopsy will be collected from the site of the implant placement for histologic evaluation

DETAILED DESCRIPTION:
10 patients will be included in this study with bilateral atrophic posterior mandible for split mouth research

. group I: prefabricated CAD-CAM allogeneic bone block sterilized with gamma rays hydrated using hyaluronic acid group II: prefabricated CAD-CAM allogeneic bone block sterilized with gamma rays hydrated using saline solution under LA mucoperiosteal flap will be elevated to expose the atrophic ridge then the prefabricated CAD-CAM allogenic block either mixed with hyaluronic acid (group I) or saline (group II) will be fixed in its position with titanium miniscrews , The block was coated with a nonporous d-PTFE membrane then closure of flap with nylon second stage: 6 months later exposure of alveolar ridge core biopsy was taken for histological study then insertion of titanium implants.

the aim of the study is to investigate the effect of hyaluronic acid on a prefabricated CAD- CAM bone blocks for ridge augmentation radiographically and histologically.

ELIGIBILITY:
Inclusion criteria:

* Patients between 40 to 65 years old.
* Posterior atrophic mandibular ridge indicated for horizontal and vertical ridge augmentation for dental implant placement.
* Good oral hygiene

Exclusion Criteria:

* Systemic diseases that affect host healing responses.
* Heavy smoking.
* Poor oral hygiene.
* Traumatic occlusion, sever para-functional habits (ex. bruxism, clenching,)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
measurement the width and the height of the alveolar ridge | 6 months
  using CBCT the width and the height will be measured with measuring tools in milimeter (mm)
the amount of new bone formation | 6 months
  core biopsy will be underwent histomorphometric analysis to determine the percentage of new bone formation (%)

SECONDARY OUTCOMES:
the sucess of dental implants | 12 months
  usingCBCT to determine the amount of marginal bone loss in (mm)

CONTACTS AND LOCATIONS:
Overall Officials: mohamed h helal, lecturer, Principal Investigator — Tanta University
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

REFERENCES:
- [Derived] Helal MH, Sheta MS, Alsherif AA, Hassan MA, Aboushelib MN, Ghouraba RF. The Effectiveness of Hyaluronic Acid on Prefabricated CAD CAM Bone Blocks for Ridge Augmentation: A Split Mouth Study. Clin Implant Dent Relat Res. 2025 Apr;27(2):e70035. doi: 10.1111/cid.70035. PMID 40231349